CLINICAL TRIAL: NCT01063283
Title: A Randomized, Open-Label, Dose Escalation Study of Bevacizumab With Ambulatory Blood Pressure Monitoring in Previously Untreated Patients With Advanced Non-squamous Non-Small Cell Lung Cancer
Brief Title: Dose Escalation of Bevacizumab With Ambulatory Blood Pressure Monitoring in Patients With Advanced Non-squamous NSCLC
Acronym: AVF4759
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-014-B
Record Dates: First submitted 2010-02-03; First posted 2010-02-05 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Advanced Non-squamous Non-Small Cell Lung Cancer
Keywords: Non-squamous Non-Small Cell Lung Cancer; Bevacizumab; Ambulatory Blood Pressure Monitoring
MeSH Terms: interventions — Pemetrexed; Carboplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): Carboplatin and Pemetrexed with Bevacizumab 7.5 mg/kg once, followed three weeks later by Carboplatin and Pemetrexed with Bevacizumab 7.5 mg/kg and bevacizumab every 3 weeks for two doses
  Interventions: Drug: Pemetrexed; Drug: Carboplatin; Drug: Bevacizumab 7.5 mg/kg
- Group B (Active Comparator): Carboplatin and Pemetrexed with Bevacizumab 7.5 mg/kg once, followed three weeks later by Carboplatin+Pemetrexed+Bevacizumab 15 mg/kg and bevacizumab every 3 weeks for two doses
  Interventions: Drug: Pemetrexed; Drug: Carboplatin; Drug: Bevacizumab 7.5 mg/kg; Drug: Bevacizumab 15 mg/kg

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed 500 mg/m^2 intravenously over 10 minutes
Drug: Carboplatin — Carboplatin at a dose calculated to produce an area under the concentration-time curve of 6 mg/ml•min intravenously over 30 minutes
Drug: Bevacizumab 7.5 mg/kg — Bevacizumab at 7.5 mg/kg intravenously over 90 minutes
Drug: Bevacizumab 15 mg/kg — Bevacizumab at 15 mg/kg intravenously over 90 minutes
  Arms: Group B

SUMMARY:
The purpose of this study is to see if higher dose of bevacizumab can be taken safely by some patients and if changes in the dose of bevacizumab have any effect on blood pressure.

DETAILED DESCRIPTION:
Carboplatin and pemetrexed are FDA approved chemotherapy agents for patients with advanced non squamous non small cell lung cancer. Bevacizumab is also FDA approved in lung cancer , and the combination of all three drugs is promising. The doctors directing this research want to learn how to better personalize drug dosing of bevacizumab by identifying people who could safely take a higher dose of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed, newly diagnosed Stage IIIB, stage IV, or recurrent non-squamous NSCLC for which they have not received chemotherapy.
* Patients must have completed radiation therapy 2 weeks prior to enrollment. Patients may have received adjuvant therapy, provided the regimen included no more than one of the study agents.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension.
* Age >18 years. •Life expectancy of greater than 4 months.
* ECOG performance status of 0 or 1
* Patients must have normal organ and marrow function
* Patients on anticoagulation are allowed.
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Disease-Specific

* Patients who have had received prior chemotherapy (in the setting of recurrent disease, other than their original adjuvant therapy)
* Patients may not be receiving any other investigational agents.
* Patients with histologic evidence of predominantly squamous lung cell cancer

  * General Medical Exclusions
* Inability to comply with study and/or follow-up procedures
* Malignancy other than superficial basal cell and superficial squamous of the skin or carcinoma in situ of the cervix within last five years

Bevacizumab-Specific Exclusions

* Inadequately controlled hypertension
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to Day 1
* History of stroke or transient ischemic attack within 6 months prior to Day 1
* Known CNS disease, except for treated brain metastasis.
* Significant vascular disease within 6 months prior to Day 1
* History of hemoptysis within 1 month prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
* History of diverticulitis, abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria as demonstrated by a UPC ratio 1.0 at screening
* Known hypersensitivity to any component of bevacizumab
* Pregnancy (positive pregnancy test) or lactation.
* Mixed tumors will be categorized by the predominant cell type unless small cell elements are present.
* Uncontrolled intercurrent illness including, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
* Any unstable condition that in the opinion of the investigator is likely to interfere with collection of accurate blood pressure measurement data .
* HIV-positive patients on combination antiretroviral therapy.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Maitland, MD., Ph.d, Principal Investigator — The University of Chicago Medical Center; Michael Maitland, MD., PhD, Principal Investigator — The University of Chicago Medical Center
Locations (3):
- United States (3):
  - The University of Chicago Medical Center, Chicago, Illinois
  - North Shore University Health System, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled patients received one cycle and those who tolerated it and had no evidence of risk for dose escalation were randomized to receive one of two treatment regimens.
Groups:
- All Participants: All participants enrolled received Carboplatin and Pemetrexed with Bevacizumab 7.5 mg/kg once during the first cycle.
- Group A: Carboplatin and Pemetrexed with Bevacizumab 7.5 mg/kg once during first cycle, followed three weeks later by Carboplatin and Pemetrexed with Bevacizumab 7.5 mg/kg and bevacizumab every 3 weeks for two doses
- Group B: Carboplatin and Pemetrexed with Bevacizumab 7.5 mg/kg once during first cycle, followed three weeks later by Carboplatin+Pemetrexed+Bevacizumab 15 mg/kg and bevacizumab every 3 weeks for two doses
Period: Cycle 1
Arm/Group | All Participants | Group A | Group B
Started | 20 | 0 | 0
Completed | 17 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Technical failure in data collection | 1 | 0 | 0
Period: Randomized Phase (Cycle 2 and Beyond)
Arm/Group | All Participants | Group A | Group B
Started | 0 | 6 | 11
Completed | 0 | 6 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients enrolled and evaluable during the randomization phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 6 | 11 | 17
Age, Continuous [Mean (Full Range); unit: years] | 53 [41 to 65] | 59 [33 to 72] | 57 [33 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 2 | 5 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-Hispanic | 4 | 4 | 8
  Black non-Hispanic | 2 | 5 | 7
  Asian | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 11 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in 24 Hour Diastolic Blood Pressure (DBP)
Description: The change for each patient was calculated as mean 24 hour DBP during cycle 2 - mean 24 hour DBP during cycle 1
Time Frame: 2 cycles
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group A | Group B
Number analyzed (Participants) | 6 | 11
mmHg | 3 (4) | 3 (10)

2. Secondary Outcome: Response Rate
Description: Percentage of patients with a complete or partial response. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 6 | 11
Participants | 3 | 2

3. Secondary Outcome: Change in Tumor Size From Baseline
Time Frame: 2 years
Population: Because the study did not meet its accrual goals, the study team did not proceed to collect this secondary outcome measure. The data were not collected and therefore are not available to report.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Progression Free Survival
Description: Time to progression or death from any cause, whichever comes first
Time Frame: 2 years
Population: as for outcome 3
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Other adverse events grade 2 or higher are reported.
Arm/Group | Group A | Group B
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/11
Other Adverse Events (participants affected / at risk) | 6/6 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=6) | Group B (N=11)
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=6) | Group B (N=11)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3
Chest pain (General disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Diaphoresis (General disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 4
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Retinal tear (Eye disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
pain (General disorders) | 1 | 4
Oral pain (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Proteinuria (Renal and urinary disorders) | 1 | 0
Swollen feet (General disorders) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Upper respiratory symptoms (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 4
Mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
white blood cell decreased (Investigations) | 0 | 1
Fatigue (General disorders) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 1
urinary tract infection (Infections and infestations) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Stroke (Nervous system disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Creatinine increased (Investigations) | 0 | 3
GERD (Gastrointestinal disorders) | 0 | 1
Intermittent periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 1
Sinus infection (Infections and infestations) | 0 | 1
Thrush (Infections and infestations) | 0 | 1
otitis externa (Infections and infestations) | 0 | 2
heart murmur (Cardiac disorders) | 0 | 1
Hepatitis (Infections and infestations) | 0 | 1

LIMITATIONS AND CAVEATS:
Recruitment was slow and the study did not meet its accrual goals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No